CLINICAL TRIAL: NCT03599570
Title: Improving HPV Vaccination Delivery in Pediatric Primary Care: The STOP-HPV Trial 2 Comparison of Performance Feedback (in the Presence of Communication Skills) and Standard of Care
Brief Title: The STOP-HPV Trial 2: Performance Feedback Intervention
Acronym: STOP-HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital of Philadelphia (Other); American Academy of Pediatrics (Other); University of Pennsylvania (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); University of Rochester (Other)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor of Pediatrics, Executive Vice-Chair and Vice-Chair for Research, Department of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R01CA202261 (NIH); R01CA202261 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-07-26 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Immunization; Vaccination
Keywords: HPV; Vaccination; Practice based intervention

STUDY DESIGN:
Intervention Model Description: A cluster RCT study design will test the impact of performance feedback to reduce missed opportunities (MOs) and raise HPV vaccine rates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Arm 1 will receive the STOP-HPV performance feedback intervention
  Interventions: Behavioral: STOP-HPV performance feedback intervention
- Control (No Intervention): Arm 2 will receive standard of care

INTERVENTIONS:
Behavioral: STOP-HPV performance feedback intervention — This intervention will be the addition of performance feedback (in the presence of communication skills).
  Arms: Intervention

SUMMARY:
Most adolescents who receive human papillomavirus (HPV) vaccine are vaccinated in pediatric practices, yet missed opportunities (MOs) for HPV vaccination occur often and lead to low HPV vaccination rates. This cluster randomized clinical trial (RCT) will test the effectiveness (and cost-effectiveness) of the addition of performance feedback (period 2) to training providers previously received on HPV vaccine communication (period 1) to reduce MOs and increase HPV vaccination rates.

DETAILED DESCRIPTION:
HPV vaccine rates remain lower than rates for other adolescent vaccines. Missed opportunities (MOs) are healthcare visits during which a patient is eligible, but does not receive a vaccine. MOs for vaccination contribute strongly to low HPV vaccination rates. This trial focuses on period 2, the addition of performance feedback in the presence of communication skills training. Arm-1 intervention study practices add performance feedback (period 2), building upon their prior training in communication skills (period 1); Arm-2 comparison study practices continue delivering standard of care. During this period, the investigators will be measuring captured opportunities - the inverse of MOs, or visits when an eligible patient receives a vaccine. Providers rarely receive feedback to track their captured opportunities, but feedback has been shown to be an effective tool. Performance feedback reports will pull from electronic health record (EHR) data, and will compare participants performance to their own previous performance and those of others. Throughout the intervention participants will also receive weekly text message mini-lessons that will remind participants of the project.

ELIGIBILITY:
Practice Inclusion Criteria:

* The practice provides HPV vaccination services to adolescents.
* The practice is part of Physician's Computer Company (PCC), Office Practicum (OP) or (a) yet-to-be selected health system(s).
* The practice has had the same EHR system in place for a year or more (with special consideration on a case by case basis if they are close to but not do not reach a year).
* The practice agrees to not participate in other HPV-related QI projects or research interventions during the study period (with special consideration on a case by case basis).

Practice Exclusion Criteria:

* The practice plans to change EHR systems in the next three years.
* The practice participated in the last year, is currently engaged in, or plans to participate in an office-based HPV-related quality improvement (QI) project or research intervention during the study period (with special consideration on a case by case basis).
* Estimated 20% or more of adolescents at the practice receive HPV vaccinations at schools or health department clinics (given standard practice and published data, the investigators expect that few to no practices will need to be excluded based on this restriction).

Patient inclusion criteria:

-All patients of participating practices (intervention and comparison) aged 11-17 years who have at least 1 visit to the practice within the past two years.

Patient exclusion criteria:

-None apart from age of patients (above).

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Change in the rate of missed vaccination opportunities among all clinicians | Monthly for Period 2 and also aggregated over the 6-month period from start date, where start date is site specific and depends on study decision on completion of training and readiness of site to proceed.
  Change in the rate of missed vaccination opportunities from baseline (period 0) through the end of period 2 among all clinicians, with a focus on the contrast between the end of period 1 and period 2.
Change in the rate of missed vaccination opportunities among consenting clinicians | Monthly for Period 2 and also aggregated over the 6-month period from start date, where start date is site specific and depends on study decision on completion of training and readiness of site to proceed.
  Change in the rate of missed vaccination opportunities from baseline (period 0) through the end of period 2 among consenting clinicians, with a focus on the contrast between periods 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- American Academy of Pediatrics, Itasca, Illinois, United States

IPD SHARING:
Plan to Share IPD: No